CLINICAL TRIAL: NCT00739349
Title: A Phase II, Multi-Center, Double-Masked, Randomized Study of NOVA22007 0.05% and 0.1% Cyclosporine Ophthalmic Cationic Emulsions Compared to Vehicle for the Treatment of the Signs and Symptoms of Dry Eye
Brief Title: NOVA22007 0.05% and 0.1% Cyclosporine Versus Vehicle for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVG08B112
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2015-06

CONDITIONS: Dry Eye
Keywords: Dry Eye; Cyclosporine
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Cyclosporine 0.05%
  Interventions: Drug: NOVA22007 ''Cyclosporine''
- 2 (Experimental): Cyclosporine 0.1%
  Interventions: Drug: NOVA22007 ''Cyclosporine''
- 3 (Placebo Comparator): vehicle/placebo
  Interventions: Drug: vehicle/placebo

INTERVENTIONS:
Drug: NOVA22007 ''Cyclosporine'' — Cyclosporine 0.05% Ophthalmic Cationic Emulsions
  Arms: 1
Drug: NOVA22007 ''Cyclosporine'' — Cyclosporine 0.1% Ophthalmic Cationic Emulsions
  Arms: 2
Drug: vehicle/placebo — vehicle/placebo
  Arms: 3

SUMMARY:
Study is to assess the safety and efficacy of NOVA22007 0.05% and 0.1% Cyclosporine Ophthalmic Cationic Emulsions QD compared to vehicle for the treatment of the signs and symptoms of dry eye after a 3 month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18 years and older
* Diagnosis of dry eye in both eyes

Exclusion Criteria:

* Contraindications to the use of the study medications
* Known allergy or sensitivity to the study medications or their components
* Female currently pregnant, nursing, or planning a pregnancy; or woman who has a positive pregnancy test
* Have participated in an investigational drug or device study within 30 days of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety and efficacy of two doses of NOVA22007 0.05% and 0.1% Cyclosporine Ophthalmic Emulsions | Approximately 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Central Maine Eye Care, PA, Lewiston, Maine, United States